CLINICAL TRIAL: NCT04742023
Title: Post-operative Complications and Graft Survival With Conventional Versus Continuous Glucose Monitoring in Patients With Diabetes Mellitus Undergoing Renal Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0066
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental)
  Interventions: Device: Continuous Glucose Monitor Application; Diagnostic Test: Finger Stick Glucose Measurement; Drug: Insulin
- Control Arm (Placebo Comparator)
  Interventions: Diagnostic Test: Finger Stick Glucose Measurement; Drug: Insulin; Device: Continuous Glucose Monitor Placebo Applied

INTERVENTIONS:
Device: Continuous Glucose Monitor Application — The Guardian™ Sensor glucose sensor is part of the Medtronic Continuous Glucose Monitoring (CGM) system. The system then uses these signals to provide sensor glucose values. Patients post-renal transplantation will have CGMs applied and values interpreted by nursing.
  Arms: Intervention Arm
Diagnostic Test: Finger Stick Glucose Measurement — Patients post-renal transplant will have finger-stick glucose measurements checked prior to meals.
Drug: Insulin — Insulin will be administered.
Device: Continuous Glucose Monitor Placebo Applied — The Guardian™ Sensor glucose sensor is part of the Medtronic Continuous Glucose Monitoring (CGM) system. The system then uses these signals to provide sensor glucose values. Patients post-renal transplantation will have CGMs applied however values will not be interpreted.
  Arms: Control Arm

SUMMARY:
This will be a prospective, randomized, single-blinded controlled trial in which the investigators evaluate post-operative serum glucose control using conventional point-of-care glucose monitoring in the morning and before meals (standard of care) versus continuous glucose monitoring using the Medtronic Guardian™ Sensor 3 continuous glucose monitor. The investigators will compare the average daily glucose level in the post-operative period (through post-operative day five) between the two arms in patients with diabetic nephropathy immediately post-renal transplant. This will serve as a pilot study to in order to power a main study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older
4. Undergoing first-time renal transplantation
5. Have a pre-existing diagnosis of Type 2 diabetes mellitus

Exclusion Criteria:

1. Age less than 18 years
2. Use of insulin pump at time of transplant
3. Insulin infusion requirement during hospitalization
4. Pregnancy or lactation
5. Known allergic reaction to Guardian™ Sensor 3 or adhesives
6. History of hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Average Daily Glucose | Postoperative day 1 - 5
  The primary outcome of this study is average daily glucose level.

SECONDARY OUTCOMES:
Number of Hyperglycemic Episodes | Postoperative days 1-5
  The number of episodes where glucose goes from <180mg/dl to ≥ 180 mg/dl.
Number of Hypoglycemic Episodes | Postoperative days 1-5
  The number of episodes where glucose levels go from > 80 mg/dl to ≤ 80 mg/dl
Total Insulin Use | Postoperative days 1-5
  The total number of insulin units used

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided